CLINICAL TRIAL: NCT01959048
Title: Efficacy and Safety of Fecal Microbiota Transplantation for Severe Clostridium Difficile Associated Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FMT for study indication has been permitted by Israeli Ministry of Health
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, STRAHILEVITZ JACOB, Senior physician, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-0676-12
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile associated disease; fecal microbiota transplantation
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fecal microbiota transplant (Experimental): fecal microbiota transplantation
  Interventions: Drug: fecal microbiota transplantation

INTERVENTIONS:
Drug: fecal microbiota transplantation

SUMMARY:
Clostridium difficile has become one of the leading causes of hospital acquired infections, and is associated with increased mortality. Patients with C. difficile associated disease (CDAD) possess deficiencies in 'normal' fecal microbial composition, most likely as a result of earlier antibiotic usage. The current standard of care treatment for severe C. difficile, which consists of antibiotics, does not restore the microbiota. Restoration of the normal colonic microbiota by fecal microbiota transplantation (FMT) may enable reversion colonic microbial population to a more 'normal'state and lead to cure.

A few patients develop severe CDAD which may be complicated by adynamic ileus, or toxic megacolon. The management in this context is based on limited data, and for some the only available option is sub-total colectomy.

Although FMT is by no means a new therapeutic modality, there is limited information on its use for the treatment of acute CDAD, including severe CDAD. Because of the high morbidity and mortality associated with treatment of patients with severe CDAD, and because the evidence supporting the current recommendations is weak and based upon the demonstration that FMT is an effective strategy to re-establish a balanced intestinal microbiota with resultant cure of recurrent CDAD, we propose to study the efficacy and safety of FMT for severe CDAD.

Patients with severe CDAD can be divided into two operational groups; those that have diarrhea and those that suffer from adynamic ileus. We propose to apply FMT through colonoscopy for all patients because current data suggest that the overall success rate of FMT for recurrent CDAD with lower gastrointestinal tract FMT was higher than FMT through the upper gastrointestinal tract. In addition, for patients with adynamic ileus and toxic megacolon (i.e., the population with the highest CDAD-associated morbidity and mortality), intra-colonic FMT administration is the preferred alternative.

DETAILED DESCRIPTION:
Screening and Consent - Index cases:

1. Hospitalized patient with the diagnosis of severe CDAD
2. At screening visit the study investigator(s) will explain the study in detail, answer any questions the candidate may have, and give the candidate a consent form to read and sign.
3. After signing the consent form, the candidate subject will be asked to provide a complete medical history and undergo a physical examination.
4. Blood will be drawn for a complete blood count (CBC) and bacterial culture
5. Stool will be collected and archived for use for further analysis as deemed necessary by the principal investigator. All analyses will be performed in an anonymous coded method, without any disclosure of the patient identifiers.

Screening and Consent - Donors:

1. Identified by recipients, generally an intimate partner or adult family member
2. Willing to donate stool
3. Exclusion criteria (per questionnaire):

   1. Had taken antibiotics within 90 days of the planned procedure
   2. Fever, diarrhea, vomiting, or any other symptoms of infection, which occurred within the two weeks prior to the day of the procedure.
   3. Known exposure to HIV or viral hepatitis (within the previous 12 months)
   4. High-risk sexual behaviors (examples: sexual contact with anyone with HIV/AIDS or hepatitis, men who have sex with men, sex for drugs or money)
   5. Use of illicit drugs
   6. Tattoo or body piercing within 6 months
   7. Incarceration within previous 12 months
   8. Known current communicable disease
   9. Risk factors for variant Creutzfeldt-Jakob disease
   10. Gastrointestinal co-morbidities
   11. History of inflammatory bowel disease
   12. History of irritable bowel syndrome, idiopathic chronic constipation, or chronic diarrhea
   13. History of gastrointestinal malignancy
   14. Recent ingestion of a potential allergen (eg, nuts) where recipient has a known allergy to this agent
   15. Systemic autoimmunity, for example, multiple sclerosis, connective tissue disease
4. Exclusion criteria (per laboratory assays):

   1. Positive HIV, hepatitis C virus, hepatitis B virus, Syphilis antibodies
   2. Stool culture positive for the enteropathogenic bacteria Salmonella, Shigella, or Campylobacter
   3. Stool stain positive for Ova and Parasites
   4. Stool positive for Giardia- and Entamoeba histolytica-specific antigens
   5. Stool positive for C. difficile toxins

Fecal Microbiota Transplantation Protocol Donor

1. Provide informed consent (laxative administration)
2. Report symptoms of infection, which occur between screening and the day of the procedure
3. Take a single dose of osmotic laxative (one tablet of "Laxadin") on the evening before the procedure
4. Provide fresh stool, at least 50 grams

Recipient 1. Provide informed consent

Fecal solution preparation

1. Universal precautions (gown, gloves, eye protection) during stool processing
2. Fresh (<6 h) donor stool specimen
3. About 50 grams of donor stool, diluted and shaken vigorously in sterile Saline 0.9% to homogeneity.
4. Filter stool through gauze if necessary to remove large debris
5. Stool suspension drawn up into 50 mL slip-tip syringes

Procedure

1. Informed consent for colonoscopy obtained including the additional theoretical risk of infection related to fecal transfusion
2. Document that examination of the colon is not adequate for cancer screening purposes (stool infusion interferes with visualization)
3. Colonoscopy performed aiming to reach the cecum with or without decompression without bowel inflation. If the cecum is not reachable the injection will be performed at the most distal site.
4. No biopsies taken
5. Upon withdrawal, injection of the fecal suspension via the biopsy channel of a colonoscope, majority into the right colon. Deliver between 300-500 ml.

Post procedure

1. Patient encouraged to retain stool (if possible) for 4 hours

Clinical and laboratory follow up

1. A blood culture will be drawn immediately following the procedure
2. Subjects will be followed during hospitalization and after discharge for at least 30 days. Data on symptoms of CDAD, on-going medical history review, physical examination, and laboratory tests as described in Table 1 will be collected.
3. Safety will be assessed by monitoring the subjects for adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders are eligible for study
2. Age 18 years and older
3. Able to provide written, informed consent
4. Confirmed diagnosis of severe CDAD as defined above

Exclusion Criteria:

(If any of the following apply, the subject MUST NOT enter the study):

1. Pregnant or lactating women
2. Need for prolonged antibiotics for other cause
3. Other known etiology for diarrhea, or clinical infection with other known enteric pathogens
4. Active, chronic conditions such as: Inflammatory bowel disease, Crohn's disease, Short bowel syndrome, Ulcerative or ischemic colitis
5. Laxatives or motility-altering drugs within 12 hours of enrolment
6. Clinically unstable. Hemodynamic instability defined as hypotension (mean arterial pressure < 60) not responsive to fluids.
7. Any condition that, in the opinion of the investigator, would preclude safe participation in the trial or compromise the quality of the data obtained.
8. Immune suppression, HIV, hematological or solid malignancy (chemotherapy in the past 3 months).
9. Prior colon surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Strahilevitz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fecal Microbiota Transplant
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 78 [71 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resolution of Severe CDAD
Description: Resolution of diarrhea, time to decrease in elevated WBC count
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
participants | 3

2. Primary Outcome: Number of Participants With Relapse of CDAD
Description: Number of Participants with evidence of relapse of C. diff. associated diarrhea
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: All Cause Mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Need for Colectomy
Description: Number of Participants who undergo colectomy due to CDAD
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Morbidity
Description: immediate colonoscopy-related complications, secondary infection
Time Frame: 1 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Arm/Group | Fecal Microbiota Transplant
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplant (N=3)
Death (Musculoskeletal and connective tissue disorders) | 1 (1) — Five days post FMT patient fell from bed and sustained fracture of femur. Was not operated and died 11 days later.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes